CLINICAL TRIAL: NCT05714241
Title: BIOmarkers and PLAtelet Function Assessment in Myocardial Ischemia and Non Obstructive Coronary Arteries Study: The BIOplatINO Study
Brief Title: BIOmarkers and PLAtelet Function Assessment in Myocardial Ischemia and Non Obstructive Coronary Arteries Study
Acronym: BIOplatINO
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, MONTONE ROCCO ANTONIO, IRCCS Researcher, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 4657
Record Dates: First submitted 2023-01-27; First posted 2023-02-06 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Ischemia With no Obstructive Coronary Artery Disease
Keywords: INOCA
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, serum, plasma, platelet, peripheral blood mononuclear cells
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ischemia with non-obstructive coronary artery disease: Patients with INOCA will be defined as those presenting with either stable, chronic symptoms (stable angina or angina equivalent) and/or signs of ischemia on noninvasive testing (i.e.: exercise stress test, stress echocardiography or nuclear imaging) undergoing elective diagnostic CAG and without obstructive coronary artery disease (defined as <50% diameter stenosis and/or fractional flow reserve [FFR]>0.80 in any major epicardial vessel).
  Interventions: Other: Data extraction; Other: Blood sampling; Other: Clinical Follow-up

INTERVENTIONS:
Other: Data extraction — After routine coronary function testing using a diagnostic pressure-temperature sensor guidewire in order to assess Coronary Flow Reserve (CFR) and the Index of Microvascular Resistance (IMR); and/or the acetylcholine (Ach) provocative test to assess the presence of coronary vasomotion disorders, patients will be stratified, accordingly to coronary function testing and Ach provocative test, in four groups/endotypes:
  1. MVA (evidence of CMD defined as any of abnormal CFR [<2.0], IMR [≥25], or microvascular spasm);
  2. VSA (CFR ≥2.0, IMR <25 and epicardial spasm);
  3. both MVA and VSA (evidence of CMD and epicardial spasm);
  4. none/non-cardiac chest pain (CFR ≥2.0 and IMR <25 and neither microvascular nor epicardial spasm).
Other: Blood sampling — At the time of this coronary angiography, arterial blood samples through the radial sheath will be collected. If collected at the time of any follow-up visit, venous blood samples will be collected by venipuncture with the same modalities to obtain whole blood, serum and plasma samples after centrifugation.
Other: Clinical Follow-up — All patients will undergo a final follow-up visit at 12 months from the date of enrollment.
  During the visit, the incidence of MACE in the past months will be investigated, the Seattle Angina Questionnaire (SAQ) will be administered and the SAQ summary score will be collected.

SUMMARY:
Ischemia with non-obstructive coronary artery disease (INOCA) identifies a significant proportion of patients presenting with signs and symptoms of myocardial ischemia with normal or near-normal coronary arteries at angiography. Initially believed a benign condition, it is now well-established that INOCA is associated with an increased risk for cardiovascular events. However, it is rarely correctly diagnosed. The identification of distinct signatures of circulating biomarkers and platelet alterations associated with the specific endotype of INOCA (Microvascular Angina [MVA]; Vasospastic Angina [VSA]; both MVA and VSA; and none) may help in the diagnosis of these patients as well as in the identification of specific pathophysiologic pathways and the development of future therapies. In addition, the identification of specific signatures may help in the prognostic stratification of INOCA patients, identifying those that may need more aggressive therapy and closer follow-up. Finally, the results deriving from this study may pave the way for a new pathophysiology-driven approach with cause-target therapies personalized for the specific mechanisms of INOCA. The BIOPLATINO study is the first study specifically designed to evaluate if there is a unique signature of circulating biomarkers and/or platelet function tests able to discriminate between the multiple pathogenetic mechanisms of INOCA as well as the different clinical courses. Furthermore, it may pave the way for the identification of specific pathophysiologic pathways of INOCA and the development of future therapies.

DETAILED DESCRIPTION:
Background

Ischemic heart diseases (IHD) still represent the leading cause of disability and mortality worldwide, with IHD and obstructive coronary artery disease (OCAD) (defined as any coronary artery stenosis ≥50%) often used as synonymous or interchangeable terms. However, a significant proportion of patients (up to 50% and particularly women) undergoing coronary angiography (CAG) because of angina and/or evidence of myocardial ischemia do not have OCAD. The term "ischemia with non-obstructive coronary artery disease" (INOCA) identifies this significant proportion of patients presenting with signs and symptoms of myocardial ischemia (e.g., angina pectoris) with normal or near-normal coronary arteries at angiography. Even if initially believed a benign condition, it is now well-established that INOCA patients are at increased risk for cardiovascular events (including acute coronary syndrome, heart failure hospitalization, stroke and repeated cardiovascular procedures). Vasomotion disorders, including microvascular angina (MVA) and/or vasospastic angina (VSA), may be particularly relevant in the pathogenesis of INOCA. Indeed, coronary vasomotion disorders can cause a relative supply-demand mismatch of myocardial blood flow and nutrients relative to their requirements, inducing myocardial ischemia that may be transient, recurrent, and/or chronic. MVA is the clinical manifestation of myocardial ischemia caused by coronary microvascular dysfunction (CMD). In this clinical entity, myocardial ischemia may result from structural remodeling of the microvasculature leading to fixed reduced microcirculatory conductance (impaired vasodilatation) and/or vasomotor disorders affecting the coronary arterioles and causing dynamic arteriolar obstruction in the presence of endothelial dysfunction and local inflammation (microvascular spasm). VSA is the clinical manifestation of myocardial ischemia caused by dynamic epicardial coronary obstruction due to epicardial artery spasm. Key subgroups of patients (endotypes) within the heterogeneous population of INOCA may be distinguished by distinct mechanisms and/or responses to medical therapy (i.e.: MVA, VSA, both MVA and VSA or none). This distinction is of mainstay importance, as the Coronary Microvascular Angina (CorMicA) trial demonstrated that a strategy of adjunctive invasive testing for disorders of coronary function linked with stratified medical therapy led to improvements in patient outcomes, including a reduction in angina severity and better quality of life. However, the specific endotype is rarely correctly diagnosed in clinical practice and, therefore, no tailored therapy is prescribed for these patients. Consequently, INOCA patients often experience recurrent angina, with hospital readmission, repeated CAG and a significant impact on quality of life and healthcare-related costs.

Platelets play pivotal roles in thrombosis and subsequent ischemic complications in patients with OCAD, and platelet activation and dysfunction have been reported also in INOCA patients. Indeed, platelets dense bodies contain adenine nucleotides (adenosine diphosphate [ADP] and adenosine triphosphate [ATP]) and serotonin which induce platelet aggregation, vasoconstriction and production of cytokines and modulators of inflammation. Moreover, healthy vascular endothelium produces potent platelet inhibitors such as nitric oxide, prostacyclin, and natural ADPase. Therefore, an imbalance in platelet activation and endothelial function, along with platelet-mediated vascular inflammation, may be relevant to the pathogenesis of INOCA. Given these diagnostic shortcomings in this evolving area of clinical research, the assessment of different circulating plasma biomarkers along with platelet function tests and their correlation with specific underlying pathophysiological mechanisms may help to identify new diagnostic and stratification tools for INOCA patients.

Hypothesis and significance

Diagnosing the precise cause, in particular, the identification of the specific endotype, is of mainstay importance in INOCA patients, given that a tailored therapy demonstrated to have a significant impact on cardiovascular and quality-of-life outcomes. Thus, the investigators hypothesized that distinct signatures of circulating biomarkers and/or platelet function may be associated with a specific endotype of INOCA. Therefore, identifying these specific signatures may help in the diagnosis of these patients as well as pave the way for the identification of specific pathophysiologic pathways and the development of future therapies. In addition, the investigators hypothesized that such specific signatures may be associated with different clinical courses at follow-up, and therefore they may help in the prognostic stratification of INOCA patients.

Thus, our hypotheses are the following:

1. that specific plasma circulating biomarkers and/or platelet function signatures could discriminate between the different endotypes of INOCA, helping to identify the underlying pathophysiological mechanisms;
2. that specific plasma circulating biomarkers and/or platelet function signatures may be associated with a worse angina status and quality of life and may be able to predict a higher rate of adverse cardiovascular events, helping in the prognostic stratification of INOCA patients and identifying those that may need more aggressive therapy and a closer follow-up.

Study design

A prospective observational pilot study.

Specific aim 1:

To evaluate the diagnostic capability of different circulating biomarkers, miRNA, platelet function tests and their combinations, in terms of sensitivity, specificity, positive predictive value (PPV) and negative predictive value (NPV) for the different endotypes of INOCA.

Specific aim 2:

To evaluate if distinct plasma circulating biomarkers and/or platelet function signatures are associated with a worse angina status and quality of life (evaluated using the Seattle Angina Questionnaire [SAQ] summary score) at 1-year follow-up in INOCA patients.

Specific Aim 3:

To evaluate if distinct circulation biomarkers and/or platelet function signatures predict worse clinical outcomes in terms of major adverse cardiovascular events (MACE) (defined as the composite of all-cause mortality, nonfatal myocardial infarction, hospitalization for angina or heart failure, stroke, and repeated CAG) at 1-year follow-up in INOCA patients.

Methods

In order to define the different endotypes of INOCA, enrolled patients will undergo or underwent a comprehensive diagnostic work-up at the time of CAG, as suggested in current guidelines and consensus, consisting of:

* Coronary function testing using a diagnostic pressure-temperature sensor guidewire in order to assess Coronary Flow Reserve (CFR) and the Index of Microvascular Resistance (IMR);
* Acetylcholine (Ach) provocative test to assess the presence of coronary vasomotion disorders;

All patients will undergo a blood sampling to assess circulating biomarkers, miRNAs expression profile and platelet function tests at the time of CAG or at the time of any follow-up visit.

Sample size calculation

To the best of our knowledge, there is no previous literature calculating sample size in a study comparing the different endotypes of INOCA. Consequently, due to the pilot nature of the study, the investigators did not perform a formal sample size calculation. However, based on data from expert consensus, the investigators assumed that a sample size of 200 patients will allow an appropriate comparison among the INOCA endotypes. Moreover, the investigators assume an enrollment rate of 50 patients/year in each participating center, thus the investigators aim at enrolling a total of 200 patients within 2 years.

Statistical analysis

Data will be reported as numbers and frequencies as for qualitative variables, whilst quantitative data will be expressed either as mean ± standard deviation (SD) or median with interquartile range (IQR). Quantitative data distribution will be assessed using the Shapiro-Wilk test. Differences between INOCA groups will be analyzed, as for qualitative data y the chi Square test. Conversely, as for quantitative data One-way ANOVA will be used for normally distributed values whereas the Kruskal-Wallis test will be performed for variables without normal distribution. The area under the curve (AUC) by receiver operating characteristics (ROC) analysis will be analysed to assess specificity, sensitivity, PPV and NPV of single-plasma biomarker, miRNAs and result of platelet function tests, as well as their combinations for different endotypes of INOCA, by using the gold-standard as reference line. Univariate and multivariate multiple linear regression will be used to evaluate the association of single-plasma biomarker, miRNAs and result of platelet function tests as well as their combinations with SAQ summary score at 1-year follow-up. Univariate and multivariate Cox regression analysis will be used to assess the relation of single-plasma biomarker, miRNAs and result of platelet function tests as well as their combinations with MACE. The analysis of MACE will consider time to first event and time to each event. A two-tailed analysis will be performed and a p value <0.05 will be considered as significant. Statistical analyses will be performed using STATA software version 16 (STATA Corp).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 18 years
* Patients diagnosed with INOCA
* Patients in therapy with acetylsalicylic acid (100 mg/die per os for more than 3 days or 250 mg intravenous in the past 3 days followed by 100 mg/die per os).

Exclusion Criteria:

* the use of thrombolytics, platelet glycoprotein (GP) IIb/IIIa blockers, oral anticoagulants, thienopyridine pretreatment, platelet counts outside the range of 125-450 10 9/l.
* comorbidities with an expected survival less than 1 year and contraindication to drugs administrated (e.g.: history of hypersensitivity to drugs administrated or its excipients, significant renal and/or hepatic disease).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with INOCA will be defined as those presenting with either stable, chronic symptoms (stable angina or angina equivalent) and/or signs of ischemia on noninvasive testing (i.e.: exercise stress test, stress echocardiography or nuclear imaging) undergoing elective diagnostic CAG and without obstructive coronary artery disease (defined as <50% diameter stenosis and/or fractional flow reserve [FFR]>0.80 in any major epicardial vessel).
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Biomarker, miRNA and platelet function assessment for the specific endotype of INOCA | Up to 30 days
  Serum levels of circulating biomarkers, miRNAs and the results of platelet function tests as well as their combinations will be analyzed to evaluate sensitivity, specificity, positive predictive value (PPV) and negative predictive value (NPV) for the specific endotype of INOCA (MVA, VSA, both MVA and VSA, or none).

SECONDARY OUTCOMES:
Biomarker, miRNA and platelet function assessment at 1 year follow up | 1 year
  Serum levels of circulating biomarkers, miRNAs and the results of platelet function tests as well as their combinations will be correlated with angina status and quality of life, evaluated using the Seattle Angina Questionnaire [SAQ] summary score, at 1-year follow-up.
Assessment of prediction model of future cardiovascular events (MACE) at 1-year follow-up. | 1 year
  Serum levels of circulating biomarkers, miRNAs, the results of platelet function tests as well as their combinations will be included in a prediction model of future cardiovascular events (MACE) at 1-year follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Rocco A Montone, MD, PhD, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (2):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Rome, Italy
- Hospital Clínic Cardiovascular Institute, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] GBD 2017 Causes of Death Collaborators. Global, regional, and national age-sex-specific mortality for 282 causes of death in 195 countries and territories, 1980-2017: a systematic analysis for the Global Burden of Disease Study 2017. Lancet. 2018 Nov 10;392(10159):1736-1788. doi: 10.1016/S0140-6736(18)32203-7. Epub 2018 Nov 8. PMID 30496103
- [Background] Kaski JC, Crea F, Gersh BJ, Camici PG. Reappraisal of Ischemic Heart Disease. Circulation. 2018 Oct 2;138(14):1463-1480. doi: 10.1161/CIRCULATIONAHA.118.031373. PMID 30354347
- [Background] Reeh J, Therming CB, Heitmann M, Hojberg S, Sorum C, Bech J, Husum D, Dominguez H, Sehestedt T, Hermann T, Hansen KW, Simonsen L, Galatius S, Prescott E. Prediction of obstructive coronary artery disease and prognosis in patients with suspected stable angina. Eur Heart J. 2019 May 7;40(18):1426-1435. doi: 10.1093/eurheartj/ehy806. PMID 30561616
- [Background] Jespersen L, Hvelplund A, Abildstrom SZ, Pedersen F, Galatius S, Madsen JK, Jorgensen E, Kelbaek H, Prescott E. Stable angina pectoris with no obstructive coronary artery disease is associated with increased risks of major adverse cardiovascular events. Eur Heart J. 2012 Mar;33(6):734-44. doi: 10.1093/eurheartj/ehr331. Epub 2011 Sep 11. PMID 21911339
- [Background] Jespersen L, Abildstrom SZ, Hvelplund A, Prescott E. Persistent angina: highly prevalent and associated with long-term anxiety, depression, low physical functioning, and quality of life in stable angina pectoris. Clin Res Cardiol. 2013 Aug;102(8):571-81. doi: 10.1007/s00392-013-0568-z. Epub 2013 May 1. PMID 23636227
- [Background] Taqueti VR, Solomon SD, Shah AM, Desai AS, Groarke JD, Osborne MT, Hainer J, Bibbo CF, Dorbala S, Blankstein R, Di Carli MF. Coronary microvascular dysfunction and future risk of heart failure with preserved ejection fraction. Eur Heart J. 2018 Mar 7;39(10):840-849. doi: 10.1093/eurheartj/ehx721. PMID 29293969
- [Background] Kunadian V, Chieffo A, Camici PG, Berry C, Escaned J, Maas AHEM, Prescott E, Karam N, Appelman Y, Fraccaro C, Louise Buchanan G, Manzo-Silberman S, Al-Lamee R, Regar E, Lansky A, Abbott JD, Badimon L, Duncker DJ, Mehran R, Capodanno D, Baumbach A. An EAPCI Expert Consensus Document on Ischaemia with Non-Obstructive Coronary Arteries in Collaboration with European Society of Cardiology Working Group on Coronary Pathophysiology & Microcirculation Endorsed by Coronary Vasomotor Disorders International Study Group. Eur Heart J. 2020 Oct 1;41(37):3504-3520. doi: 10.1093/eurheartj/ehaa503. PMID 32626906
- [Background] Ford TJ, Ong P, Sechtem U, Beltrame J, Camici PG, Crea F, Kaski JC, Bairey Merz CN, Pepine CJ, Shimokawa H, Berry C; COVADIS Study Group. Assessment of Vascular Dysfunction in Patients Without Obstructive Coronary Artery Disease: Why, How, and When. JACC Cardiovasc Interv. 2020 Aug 24;13(16):1847-1864. doi: 10.1016/j.jcin.2020.05.052. PMID 32819476
- [Background] Camici PG, Crea F. Coronary microvascular dysfunction. N Engl J Med. 2007 Feb 22;356(8):830-40. doi: 10.1056/NEJMra061889. No abstract available. PMID 17314342
- [Background] Crea F, Camici PG, Bairey Merz CN. Coronary microvascular dysfunction: an update. Eur Heart J. 2014 May;35(17):1101-11. doi: 10.1093/eurheartj/eht513. Epub 2013 Dec 23. PMID 24366916
- [Background] Del Buono MG, Montone RA, Camilli M, Carbone S, Narula J, Lavie CJ, Niccoli G, Crea F. Coronary Microvascular Dysfunction Across the Spectrum of Cardiovascular Diseases: JACC State-of-the-Art Review. J Am Coll Cardiol. 2021 Sep 28;78(13):1352-1371. doi: 10.1016/j.jacc.2021.07.042. PMID 34556322
- [Background] Maseri A. Louis F. Bishop lecture. Role of coronary artery spasm in symptomatic and silent myocardial ischemia. J Am Coll Cardiol. 1987 Feb;9(2):249-62. doi: 10.1016/s0735-1097(87)80372-8. PMID 3543091
- [Background] Ford TJ, Stanley B, Good R, Rocchiccioli P, McEntegart M, Watkins S, Eteiba H, Shaukat A, Lindsay M, Robertson K, Hood S, McGeoch R, McDade R, Yii E, Sidik N, McCartney P, Corcoran D, Collison D, Rush C, McConnachie A, Touyz RM, Oldroyd KG, Berry C. Stratified Medical Therapy Using Invasive Coronary Function Testing in Angina: The CorMicA Trial. J Am Coll Cardiol. 2018 Dec 11;72(23 Pt A):2841-2855. doi: 10.1016/j.jacc.2018.09.006. Epub 2018 Sep 25. PMID 30266608
- [Background] Ford TJ, Stanley B, Sidik N, Good R, Rocchiccioli P, McEntegart M, Watkins S, Eteiba H, Shaukat A, Lindsay M, Robertson K, Hood S, McGeoch R, McDade R, Yii E, McCartney P, Corcoran D, Collison D, Rush C, Sattar N, McConnachie A, Touyz RM, Oldroyd KG, Berry C. 1-Year Outcomes of Angina Management Guided by Invasive Coronary Function Testing (CorMicA). JACC Cardiovasc Interv. 2020 Jan 13;13(1):33-45. doi: 10.1016/j.jcin.2019.11.001. Epub 2019 Nov 11. PMID 31709984
- [Background] Bairey Merz CN, Pepine CJ, Walsh MN, Fleg JL. Ischemia and No Obstructive Coronary Artery Disease (INOCA): Developing Evidence-Based Therapies and Research Agenda for the Next Decade. Circulation. 2017 Mar 14;135(11):1075-1092. doi: 10.1161/CIRCULATIONAHA.116.024534. PMID 28289007
- [Background] Gurbel PA, Bliden KP, Hayes KM, Tantry U. Platelet activation in myocardial ischemic syndromes. Expert Rev Cardiovasc Ther. 2004 Jul;2(4):535-45. doi: 10.1586/14779072.2.4.535. PMID 15225113
- [Background] Choi JL, Li S, Han JY. Platelet function tests: a review of progresses in clinical application. Biomed Res Int. 2014;2014:456569. doi: 10.1155/2014/456569. Epub 2014 May 8. PMID 24895576
- [Background] Lanza GA, Andreotti F, Sestito A, Sciahbasi A, Crea F, Maseri A. Platelet aggregability in cardiac syndrome X. Eur Heart J. 2001 Oct;22(20):1924-30. doi: 10.1053/euhj.2001.2624. PMID 11601836
- [Background] Chan PS, Jones PG, Arnold SA, Spertus JA. Development and validation of a short version of the Seattle angina questionnaire. Circ Cardiovasc Qual Outcomes. 2014 Sep;7(5):640-7. doi: 10.1161/CIRCOUTCOMES.114.000967. Epub 2014 Sep 2. PMID 25185249
- [Background] Knuuti J, Wijns W, Saraste A, Capodanno D, Barbato E, Funck-Brentano C, Prescott E, Storey RF, Deaton C, Cuisset T, Agewall S, Dickstein K, Edvardsen T, Escaned J, Gersh BJ, Svitil P, Gilard M, Hasdai D, Hatala R, Mahfoud F, Masip J, Muneretto C, Valgimigli M, Achenbach S, Bax JJ; ESC Scientific Document Group. 2019 ESC Guidelines for the diagnosis and management of chronic coronary syndromes. Eur Heart J. 2020 Jan 14;41(3):407-477. doi: 10.1093/eurheartj/ehz425. No abstract available. PMID 31504439